CLINICAL TRIAL: NCT03574233
Title: Ultrasonography Guided Weaning Protocol Development to Predict Successful Weaning
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2018-0357
Record Dates: First submitted 2018-06-03; First posted 2018-06-29 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Mechanical Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients who are ready to wean ventilator off

SUMMARY:
The investigators aimed to develop integrated ultrasound guided mechanical weaning protocol in critically ill patients. The analysis will be taken (1) just before the spontaneous breathing trial in enrolled patients with mechanical ventilation and (2) in patients with tracheostomy who fail ventilator off.

DETAILED DESCRIPTION:
Prolonged mechanical ventilation is associated with higher ventilator-associated pneumonia and ventilator-associated lung injury, longer intensive care unit and hospital days, increased mortality, and higher medical costs. However, some patients are difficult to wean from invasive mechanical ventilation. Typically, the difficulty in transitioning patients to spontaneous breathing may be categorized as simple transition, difficult transition, and prolonged transition.

There are a lot of predictors for weaning failure such as cardiac dysfunction, increased respiratory rate, diaphragm dysfunction, rapid shallow breathing index and so on. However, weaning failure involves complicated mechanisms that are not solved by one cause. Recently, P. Mayo published a review paper on ultrasonography evaluation during the weaning process. The investigators need to pay attention to this paper. While lots of previous predictors cannot explain the reason, ultrasound evaluation is a process of finding the cause as well as prediction for weaning failure. However, The investigators need a more practical and standardized ultrasound protocols for how to wean invasive mechanical ventilation. "Ultrasonographic mechanical weaning protocol" should not comprise just one indicator, but include various indicators such as upper airway stenosis, heart function, the status of the lung and pleura, diaphragmatic function, Etc. This integrated ultrasound protocol will help in successful weaning of invasive mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

1. Invasive mechanical ventilation > 24 hours
2. Eligibility to weaning from mechanical ventilation

Exclusion Criteria:

1. Age < 18 years old
2. Severe skin lesions or infections that cannot perform ultrasound
3. Severe subcutaneous emphysema that cannot perform ultrasound
4. Patients who completed "Do-not-resuscitation" consents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mechanically ventilation participants in a mixed intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2019-05-30 (Estimated); Study Completion 2019-05-30 (Estimated)

PRIMARY OUTCOMES:
Investigation of ultrasound indices associated with the success or failure of mechanical ventilation weaning | within 48 hours
  * Weaning success: stable without mechanical ventilator support during more than 48 hours
  * Weaning failure: unstable without mechanical ventilator support within 48 hours A) Type I respiratory failure: high flow oxygen support B) Type II respiratory failure: non-invasive ventilatory support C) Reintubation

SECONDARY OUTCOMES:
A) In-ICU mortality | 90 days after Ultrasonography
B) In-hospital mortality | 90 days after Ultrasonography
C) Ventilator free day | 90 days after Ultrasonography
D) ICU free day | 90 days after Ultrasonography

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided